CLINICAL TRIAL: NCT05269823
Title: Topical Ice-therapy for Pain Modulation During Intravitreal Injections: A Prospective Randomized Control Trial
Brief Title: Topical Ice-therapy for Intravitreal Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OPH-2022-30605
Record Dates: First submitted 2022-01-16; First posted 2022-03-08 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Anesthesia; Hypothermia; Injection Site Irritation
MeSH Terms: conditions — Hypothermia | interventions — Ice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ice-therapy (Active Comparator): Ice therapy will be provided prior to the provision of the intravitreal injection
  Interventions: Other: Ice-therapy
- No Ice-therapy (Placebo Comparator): No ice therapy will be provided prior to the provision of the intravitreal injection
  Interventions: Other: No Ice-therapy

INTERVENTIONS:
Other: Ice-therapy — Ice therapy will be provided prior to intravitreal injection provision
  Arms: Ice-therapy
Other: No Ice-therapy — No additional intervention (i.e.) ice therapy will be provided prior to intravitreal injection provision
  Arms: No Ice-therapy

SUMMARY:
Purpose: To examine the difference in patient's pain experience in the setting of intravitreal anti-VEGF injections with pretreatment of topical ice-therapy compared with no-ice.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 or older evaluated by a single retina specialist at the University of Minnesota Department of Ophthalmology with a clinical indication necessitating an anti-VEGF intravitreal injection

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Discomfort assessed by the visual analog scale | This will be assessed at five minutes after the conclusion of the intravitreal injection
  This primary outcome measure will be surveyed using a visual analog scale to quantify discomfort from a numerical level of one to ten. A self reported rating of one represents the lowest self-reported subjective rating attributed to discomfort, while a rating of ten signifies the maximum self-reported subjective rating attributed to discomfort.
Itching assessed by the visual analog scale | This will be assessed at five minutes after the conclusion of the intravitreal injection
  This primary outcome measure will be surveyed using a visual analog scale to quantify discomfort from a numerical level of one to ten. A self reported rating of one represents the lowest self-reported subjective rating attributed to itching, while a rating of ten signifies the maximum self-reported subjective rating attributed to itching.
Burning assessed by the visual analog scale | This will be assessed at five minutes after the conclusion of the intravitreal injection
  This primary outcome measure will be surveyed using a visual analog scale to quantify discomfort from a numerical level of one to ten. A self reported rating of one represents the lowest self-reported subjective rating attributed to burning, while a rating of ten signifies the maximum self-reported subjective rating attributed to burning.
Overall Pain assessed by the visual analog scale | This will be assessed at five minutes after the conclusion of the intravitreal injection
  This primary outcome measure will be surveyed using a visual analog scale to quantify discomfort from a numerical level of one to ten. A self reported rating of one represents the lowest self-reported subjective rating attributed to overall pain, while a rating of ten signifies the maximum self-reported subjective rating attributed to overall pain.
Overall Tolerability assessed by the visual analog scale | This will be assessed at five minutes after the conclusion of the intravitreal injection
  This primary outcome measure will be surveyed using a visual analog scale to quantify discomfort from a numerical level of one to ten. A self reported rating of one represents the lowest self-reported subjective rating attributed to overall tolerability, while a rating of ten signifies the maximum self-reported subjective rating attributed to overall tolerability.

SECONDARY OUTCOMES:
Discomfort assessed by the visual analog scale | This will be assessed at 24-hours after the conclusion of the intravitreal injection
  This primary outcome measure will be surveyed using a visual analog scale to quantify discomfort from a numerical level of one to ten. A self reported rating of one represents the lowest self-reported subjective rating attributed to discomfort, while a rating of ten signifies the maximum self-reported subjective rating attributed to discomfort.
Itching assessed by the visual analog scale | This will be assessed at 24-hours after the conclusion of the intravitreal injection
  This primary outcome measure will be surveyed using a visual analog scale to quantify discomfort from a numerical level of one to ten. A self reported rating of one represents the lowest self-reported subjective rating attributed to itching, while a rating of ten signifies the maximum self-reported subjective rating attributed to itching.
Burning assessed by the visual analog scale | This will be assessed at 24-hours after the conclusion of the intravitreal injection
  This primary outcome measure will be surveyed using a visual analog scale to quantify discomfort from a numerical level of one to ten. A self reported rating of one represents the lowest self-reported subjective rating attributed to burning, while a rating of ten signifies the maximum self-reported subjective rating attributed to burning.
Overall Pain assessed by the visual analog scale | This will be assessed at 24-hours after the conclusion of the intravitreal injection
  This primary outcome measure will be surveyed using a visual analog scale to quantify discomfort from a numerical level of one to ten. A self reported rating of one represents the lowest self-reported subjective rating attributed to overall pain, while a rating of ten signifies the maximum self-reported subjective rating attributed to overall pain.
Overall Tolerability assessed by the visual analog scale | This will be assessed at 24-hours after the conclusion of the intravitreal injection
  This primary outcome measure will be surveyed using a visual analog scale to quantify discomfort from a numerical level of one to ten. A self reported rating of one represents the lowest self-reported subjective rating attributed to overall tolerability, while a rating of ten signifies the maximum self-reported subjective rating attributed to overall tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Jade Moon, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided